CLINICAL TRIAL: NCT07074418
Title: Effect of Empagliflozin in Patients With eGFR Between 10 and 20 ml/Min/1.73m2 - EMPA [10-20]
Brief Title: Effect of Empagliflozin in Patients With eGFR Between 10 and 20 ml/Min/1.73m2
Acronym: EMPA[10-20]
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 23-PP-12
Record Dates: First submitted 2025-06-30; First posted 2025-07-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease; Nephrology; eGFR
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo-controlled, cross over
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): empaglifozine 10mg / wash-out / matching placebo
  Interventions: Drug: Empagliflozin 10 MG then Placebo
- Group 2 (Active Comparator): matching placebo / wash-out / empaglifozine 10mg
  Interventions: Drug: Placebo then Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG then Placebo — Taking Empagliflozin first
  Other Names: EMPAGLIFLOZIN or iSGLT2
  Arms: Group 1
Drug: Placebo then Empagliflozin 10 MG — Taking the Empagliflozin in second
  Other Names: EMPAGLIFLOZIN or iSGLT2
  Arms: Group 2

SUMMARY:
The proximal tubule remains the main site for sodium reabsorption in patients with advanced renal failure. The investigators therefore hypothesize that SGLT2i should still exert a significant natriuretic effect in patients with eGFR below 20 ml/min/1.73m2, and therefore should still decrease proteinuria with a potential renal protective effect.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetics,
* age between 18 and 80 years,
* RAS blockade at maximal tolerated dosage for 1 month,
* eGFR (CKD-EPI) between 10 and 20 ml/min/1.73m2,
* UACR > 300mg/g creatinine and UPCR > 500mg/g creatinine,
* office systolic blood pressure > 110 mmHg,
* stable dosage of antihypertensive drugs and diuretics for 1 month.

Exclusion Criteria:

* any medical condition that, in the opinion of the investigator makes the participant not suitable for inclusion,
* history of ketoacidosis in the past while on empagliflozin or any other SGLT2i class drugs,
* participation in another clinical study with an investigational medicinal product (IMP) administered during the month before screening,
* known hypersensitivity or intolerance to empagliflozin or any of the excipients of the product,
* judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements,
* no social insurance,
* unwilling to give informed consent, vulnerable persons (minors, adults under guardianship or trusteeship, pregnant women, persons deprived of their liberty, persons unable to speak French).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Anti-proteinuric effect | 20 months
  Changes in mean UACR on spot morning urine samples between 2 days running at baseline and 2 days running at the end of each 6-week treatment period (empagliflozin 10 mg/d and matching placebo).
  To show that in type 2 diabetic patients with eGFR between 10 and 20 ml/min/1.73m2, SGLT2i exerts a clinically significant anti-proteinuric effect.

SECONDARY OUTCOMES:
Body weight effect | 20 months
  Changes in body weight between baseline and at the end of each 6-week treatment period (empagliflozin 10 mg/d and matching placebo.
  To show that in type 2 diabetic patients with eGFR between 10 and 20 ml/min/1.73m2, empagliflozin acutely decreases body weight.
Urinary sodium effect | 20 months
  To show that in type 2 diabetic patients with eGFR between 10 and 20 ml/min/1.73m2, empagliflozin:
  increases urinary sodium excretion. Changes in mean UPCR on spot morning urine samples between 2 days running at baseline and 2 days running at the end of each 6-week treatment period (empagliflozin 10 mg/d and matching placebo).
Urinary volume effect | 20 months
  To show that in type 2 diabetic patients with eGFR between 10 and 20 ml/min/1.73m2, empagliflozin:
  increases urinary volume. Changes in mean 24-hour urinary.
Blood pressure effect | 20 months
  To show that in type 2 diabetic patients with eGFR between 10 and 20 ml/min/1.73m2, empagliflozin: decreases ambulatory blood pressure.
  Changes in mean ambulatory systolic blood pressure between 3 days running baseline and 3 days running at the end of each 6-week treatment period (empagliflozin 10 mg/d and matching placebo).
eGFR effect by good profile | 20 months
  To show that in type 2 diabetic patients with eGFR between 10 and 20 ml/min/1.73m2, empagliflozin has a good safety profile (no acute kidney injury or hyperkalaemia > 5.5 mmol/L or acidosis (serum bicarbonate <23 mmol/L)),
eGFR effect by levels | 20 months
  Changes in eGFR levels between baseline and every week during each 6-week treatment period (empagliflozin 10 mg/d and matching placebo).
eGFR effect by serum potassium | 20 months
  Changes in serum potassium levels between baseline and every week during each 6-week treatment period (empagliflozin 10 mg/d and matching placebo).
eGFR effect by serum bicarbonate | 20 months
  Changes in serum bicarbonate levels between baseline and every week during each 6-week treatment period (empagliflozin 10 mg/d and matching placebo).
eGFR effect by albuminuria | 20 months
  Changes in mean 24-hour albuminuria between 3 days running urinary collections at baseline and after starting each treatment period (empagliflozin 10 mg/d and matching placebo).
Effect on HbA1c | 20 months
  To show that in type 2 diabetic patients with eGFR between 10 and 20 ml/min/1.73m2, empagliflozin has no significant effect on HbA1c.
  Changes in HbA1C between baseline and at the end of each 6-week treatment period (empagliflozin 10 mg/d and matching placebo).
Magnitude of eGFR by TEAEs | 20 months
  Describe the magnitude of eGFR decrease following empagliflozin or placebo treatments with the description of treatment emergent adverse events (TEAEs).
Magnitude of eGFR by SAEs | 20 months
  Describe the magnitude of eGFR decrease following empagliflozin or placebo treatments with the description of serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent ESNAULT, MD-PHD, Principal Investigator — CHU NICE
Locations (1):
- CHU Nice - Hôpital Pasteur 2, Nice, Alpes-Maritimes, France